CLINICAL TRIAL: NCT04404374
Title: Efficacy of a New-generation Platelet-rich Fibrin vs. Enamel Matrix Derivatives in the Treatment of Periodontal Intrabony Defects : a Randomized Clinical Trial
Brief Title: Treatment of Periodontal Intrabony Defects With A-PRF+ or EMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Boroka Csifo-Nagy, Assistant Professor, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SE TUKEB: 254/2017
Record Dates: First submitted 2020-05-19; First posted 2020-05-27 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Periodontal Diseases
Keywords: Intrabony Defects; New-Generation Platelet-Rich Fibrin; Enamel Matrix Derivatives; Periodontal Regeneration; EMD; A-PRF+; Advanced Platelet-Rich Fibrin
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A-PRF (Active Comparator): Advanced Platelet-Rich Fibrin
  Interventions: Procedure: A-PRF/EMD
- EMD (Active Comparator): Enamel Matrix Derivatives
  Interventions: Procedure: A-PRF/EMD

INTERVENTIONS:
Procedure: A-PRF/EMD — Comparing healing effect of an autologous and a xenogenic product

SUMMARY:
The aim of this randomized clinical trial was to clinically evaluate and compare the healing of intrabony defects after treatment with advanced platelet-rich fibrin (A-PRF+) to enamel matrix derivatives (EMD) in periodontitis patients.

DETAILED DESCRIPTION:
Thirty (30) intrabony defects of 18 patients (9 males, 9 females) were randomly divided in two treatment groups: test (n = 15) and control (n = 15). The intrabony defects were filled with A-PRF+ (n=15) in the test group, respectively with EMD in the control group, and fixed with sutures to ensure wound closure and stability.

ELIGIBILITY:
Inclusion Criteria:

* no systemic diseases that could influence the outcome of the therapy, a good level of oral hygiene, he presence of a 2-, 3-, or combined 2-3-wall intrabony defect with a defect angle of 20-40 (+/- 5) degrees, with a minimum PPD of 6 mm and intrabony component of a minimum 4 mm as detected on radiographs, no smoking

Exclusion Criteria:

* systemic diseases that could influence the outcome of the therapy, poor oral hygiene, smoking, horizontal bone loss

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Periodontal clinical parameters - to determine the clinical attachment level (CAL) | Change from baseline after 6 month and after 12 month
  With a calibrated periodontal probe we are examining the changes of periodontal probing depth (PPD) and gingival recession (GR) after surgical procedure in mm, the two parameters are used to determine the clinical attachment level (CAL).
Periodontal clinical parameters | Change from baseline after 6 month and after 12 month
  With a calibrated periodontal probe we are examining the changes of periodontal probing depth (PPD) and gingival recession (GR) after surgical procedure in mm, the two parameters are used to determine the clinical attachment level (CAL).

CONTACTS AND LOCATIONS:
Overall Officials: Ferenc Dr.Dőri, professor, Study Director — Semmelweis University
Locations (1):
- Semmelweis University, Department of Periodontology, Budapest, Hungary

REFERENCES:
- [Derived] Csifo-Nagy BK, Solyom E, Bognar VL, Nevelits A, Dori F. Efficacy of a new-generation platelet-rich fibrin in the treatment of periodontal intrabony defects: a randomized clinical trial. BMC Oral Health. 2021 Nov 15;21(1):580. doi: 10.1186/s12903-021-01925-1. PMID 34781955